CLINICAL TRIAL: NCT04306224
Title: A First-in-Human, Open-Label, Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of IMC-002 in Subjects With Metastatic or Locally Advanced Solid Tumors and Relapsed or Refractory Lymphomas
Brief Title: A Study of IMC-002 in Subjects With Metastatic or Locally Advanced Solid Tumors and Relapsed or Refractory Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneOncia Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMC-002-101
Record Dates: First submitted 2020-03-06; First posted 2020-03-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor; Lymphoma
Keywords: IMC-002; Phase I; CD47; SIRPα
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: Dose escalation will consist of two distinct sub-parts (1A and 1B).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMC-002 (Experimental): Dose escalation will follow the traditional 3+3 design.
  Interventions: Biological: IMC-002

INTERVENTIONS:
Biological: IMC-002 — IMC-002 blocks the interaction between CD47 and SIRPα.

SUMMARY:
This is the first-in-human, Phase I, open-label, multiple-ascending dose study to investigate the safety, tolerability, PK, PharmDyn, and clinical activity of IMC-002 in subjects with metastatic or locally advanced solid tumors and relapsed or refractory lymphomas.

Male or female subjects 18 years and older with metastatic or locally advanced solid tumors and relapsed or refractory lymphomas will be included in the study if they meet all the inclusion criteria and none of the exclusion criteria.

The study will consist of 2 parts:

Part 1: Dose Escalation Part 2: Expansion Cohorts

DETAILED DESCRIPTION:
Part 1: Dose Escalation

Part 2: Expansion Cohort The study may be amended in the future to include expansion cohorts in selected tumor types to further evaluate extended safety of IMC-002 at recommended Phase 2 dose in that tumor type. Sample size in the Dose Expansion part will be determined when the study is amended to include the expansion cohorts.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible to be included in the study only if all of the following criteria apply:

1. Signed informed consent form (ICF)
2. Adult (18 years or older)
3. Histologically or cytologically proven metastatic or locally advanced solid tumors and relapsed or refractory lymphomas, for which no standard therapy known to prolong survival exists or have relapsed/refractory/PD following the last line of treatment
4. Solid tumors must be measurable with at least 1 unidimensional measurable lesion by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Lymphomas must have at least 1 measurable lesion according to the Lugano criteria with the Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) modification
5. Availability of tumor archival material or fresh biopsies for measurement of CD47
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at Screening and an estimated life expectancy of at least 3 months
7. Adequate hematologic function, hepatic function, and renal function

Exclusion Criteria

Subjects are excluded from the study if any of the following criteria apply:

1. Treatment with nonpermitted drugs (within 28 days before Day 1).
2. Prior treatment with a CD47 or SIRPα targeting agent
3. Concurrent anticancer treatments within 28 days before Day 1/first study treatment administration
4. Major surgery or significant traumatic injury within 6 weeks prior to Screening or planned major surgery during the study period
5. Previous malignant disease other than the target malignancy for this study, except adequately treated Stage I or II cancers from which the subject is currently in complete remission per the Investigator's clinical judgment
6. Primary central nervous system (CNS) disease or leptomeningeal disease; known CNS metastases unless treated
7. Comorbidities/medical history of any significant diseases that in the judgment of the Investigator would make the subject inappropriate for this study
8. Active infection requiring systemic therapy within 14 days before Day 1
9. Persisting toxicities Grade > 1 NCI-CTCAE Version 5.0 related to prior anticancer treatment
10. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities (DLT) | For 28 days
Incidence and severity of adverse events (AEs) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: HEUNG TAE KIM, Study Director — ImmuneOncia Therapeutics Inc.
Locations (4):
- United States (3):
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No